CLINICAL TRIAL: NCT04297865
Title: A Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Phase 1 Clinical Trial to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of CJ-15314 Phosphate in Healthy Male Subjects
Brief Title: Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of CJ-15314 Phosphate in Healthy Male Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CJ_JSI_101
Record Dates: First submitted 2020-02-21; First posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- A dose as CJ-15314 or placebo (Experimental): Oral administration of A as CJ-15314 or placebo once a day
  Interventions: Drug: A dose as CJ-15314; Drug: Placebo
- B dose as CJ-15314 or placebo (Experimental): Oral administration of B as CJ-15314 or placebo once a day
  Interventions: Drug: B dose as CJ-15314; Drug: Placebo
- C dose as CJ-15314 or placebo (Experimental): Oral administration of C as CJ-15314 or placebo once a day and once daily for 7 days
  Interventions: Drug: C dose as CJ-15314; Drug: Placebo
- D dose as CJ-15314 or placebo (Experimental): Oral administration of D as CJ-15314 or placebo once a day and once daily for 7 days
  Interventions: Drug: D dose as CJ-15314; Drug: Placebo
- E dose as CJ-15314 or placebo (Experimental): Oral administration of E as CJ-15314 or placebo once a day and once daily for 7 days
  Interventions: Drug: E dose as CJ-15314; Drug: Placebo
- F dose as CJ-15314 or placebo (Experimental): Oral administration of F as CJ-15314 or placebo once a day and once daily for 7 days
  Interventions: Drug: F dose as CJ-15314; Drug: Placebo

INTERVENTIONS:
Drug: A dose as CJ-15314 — A dose as CJ-15314, 1 capsule
  Arms: A dose as CJ-15314 or placebo
Drug: B dose as CJ-15314 — B dose as CJ-15314, 1 capsule
  Arms: B dose as CJ-15314 or placebo
Drug: C dose as CJ-15314 — C dose as CJ-15314, 1 capsule
  Arms: C dose as CJ-15314 or placebo
Drug: D dose as CJ-15314 — D dose as CJ-15314, 2 capsules
  Arms: D dose as CJ-15314 or placebo
Drug: E dose as CJ-15314 — E dose as CJ-15314, 1 capsule
  Arms: E dose as CJ-15314 or placebo
Drug: F dose as CJ-15314 — F dose as CJ-15314, 2 capsules
  Arms: F dose as CJ-15314 or placebo
Drug: Placebo — Placebo, 1 capsule
  Arms: A dose as CJ-15314 or placebo
Drug: Placebo — Placebo, 1 capsule
  Arms: B dose as CJ-15314 or placebo
Drug: Placebo — Placebo, 1 capsule
  Arms: C dose as CJ-15314 or placebo
Drug: Placebo — Placebo, 2 capsules
  Arms: D dose as CJ-15314 or placebo
Drug: Placebo — Placebo, 1 capsule
  Arms: E dose as CJ-15314 or placebo
Drug: Placebo — Placebo, 2 capsules
  Arms: F dose as CJ-15314 or placebo

SUMMARY:
This study aims to evaluate safety, tolerability, pharmacokinetics and pharmacodynamics of CJ-15314 phosphate in healthy male subjects.

DETAILED DESCRIPTION:
* To evaluate the safety, tolerability and pharmacokinetics of single or multiple dose of CJ-15314 phosphate in healthy male subjects
* To explore the pharmacodynamics of single or multiple dose of CJ-15314 phosphate in healthy male subjects
* To explore the pharmacokinetics of CJ-15314 Phosphate active metabolites of single or multiple dose of CJ-15314 phosphate in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male adults aged 19 to 55 years (inclusive) at the time of signing the informed consent form.
* Body mass index (BMI) ≥ 18.0 and ≤ 30.0 kg/m^2 with a body weight ≥ 50.0 kg and ≤ 90.0 kg at screening.

  ☞ BMI (kg/m^2) = weight (kg) / {height (m)}^2
* Decides to participate voluntarily in the study after being fully informed of and understanding the study completely, and provides his written informed consent prior to screening procedure.
* Determined eligible for this study in the opinion of the investigator based on the results of vital signs, physical examination, 12-lead electrocardiogram, clinical laboratory tests, and medical interview drug screening test.

Exclusion Criteria:

* Has a history or current evidence of clinically significant disorder of hepatic, renal, nervous, respiratory, endocrine, hemato-oncologic, cardiovascular, urinary, and/or psychiatric system.
* Has a history or current evidence of gastrointestinal disease that may affect the safety and PD assessment of IP or a history of gastrointestinal surgery (except for simple appendectomy or herniotomy).
* Has rheumatoid arthritis or has a history.
* Has symptomatic herpes simplex or herpes zoster or has a history within 3 months prior to the scheduled first dose.
* Has live vaccine dose within 3 months prior to the scheduled first dose or expects to receive live vaccine during the clinical trial period.
* Has a history or current evidence of clinically significant hypersensitivity to drugs containing any ingredient of Janus kinase inhibitor and other drugs.
* Has a positive result on serology tests (for hepatitis B, hepatitis C and human immunodeficiency virus [HIV]) during screening test.
* Has abnormalities one or more of the following during screening test: AST [GOT] or ALT [GPT] > 1.5 X upper limit of normal (ULN), Creatinine > upper limit of normal (ULN), ANC < 2,000/uL, Hb <12.5 g/dL, Platelet < 150,000/uL, QTc interval at 12-lead electrocardiogram > 450 msec
* Systolic blood pressure (SBP) < 90 mmHg or > 140 mmHg, diastolic blood pressure (DBP) < 50 mmHg or > 95 mm Hg, or pulse rate (PR) < 45 beats/min or > 100 beats/min on vital signs measured in sitting position after taking a rest for at least 5 minutes during screening test.
* Has a history of drug abuse or has a positive response to drug abuse on urine drug screening test.
* Has taken any prescription drugs or herbal medicine within 2 weeks prior to the expected date of first dose, or has taken or is expected to take any over-the-counter (OTC) drug, health functional food or vitamin preparation within 1 week prior to the expected date of the first dose (However, can participate in the study if otherwise eligible in the judgment of the investigator).
* Has participated in any other clinical study or bioequivalence study and received IPs within 6 months prior to the scheduled first dose.
* Has donated whole blood within 2 months prior to the scheduled first dose, or has donated blood components or received transfusion within a month prior to the scheduled first dose.
* Has a history of excessive smoking (> 10 cigarettes/day) within 3 months prior to the scheduled first dose or confirmed as positive for cotinine on urine drug screening test.
* Excessive caffeine intake (> 5 units/day), continued use of alcohol (> 21 units/week, 1 unit = 10 g of pure alcohol), or unable to stop drinking during hospitalization period.
* Unable to avoid caffeine-containing foods (e.g., coffee, tea [black tea, green tea, etc.], soda, coffee-flavored milk, and nutritive tonic drink) during the period from 24 hrs before hospitalization to discharge.
* Unable to use a medically acceptable contraceptive method throughout the study.

  ► Medically acceptable contraceptive methods include:
  1. Use of intrauterine device with a proven birth control failure rate by the spouse (or partner)
  2. Simultaneous use of (male or female) barrier method and spermicide
  3. Surgical sterilization of the subject or his partner (e.g., vasectomy, salpingectomy, tubal ligation, or hysterectomy)
* Determined ineligible for study participation by the investigator for other reasons such as clinical laboratory abnormalities.

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2020-02-24 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Cmax of single dose of CJ-15314 | Up to 72 hours
Tmax of single dose of CJ-15314 | Up to 72 hours
AUClast of single dose of CJ-15314 | Up to 72 hours
AUCinf of single dose of CJ-15314 | Up to 72 hours
t1/2 of single dose of CJ-15314 | Up to 72 hours
λz of single dose of CJ-15314 | Up to 72 hours
CL/F of single dose of CJ-15314 | Up to 72 hours
Vd/F of single dose of CJ-15314 | Up to 72 hours
Ae of single dose of CJ-15314 | Up to 72 hours
fe of single dose of CJ-15314 | Up to 72 hours
CLR of single dose of CJ-15314 | Up to 72 hours
Cmax,ss of multiple doses of CJ-15314 | Up to 72 hours
Cmin,ss of multiple doses of CJ-15314 | Up to 72 hours
Cav,ss of multiple doses of CJ-15314 | Up to 72 hours
Tmax,ss of multiple doses of CJ-15314 | Up to 72 hours
AUCtau,ss of multiple doses of CJ-15314 | Up to 72 hours
t1/2 of multiple doses of CJ-15314 | Up to 72 hours
PTF of multiple doses of CJ-15314 | Up to 72 hours
Ra of multiple doses of CJ-15314 | Up to 72 hours
Ae of multiple doses of CJ-15314 | Up to 72 hours
fe of multiple doses of CJ-15314 | Up to 72 hours
CLR of multiple doses of CJ-15314 | Up to 72 hours

SECONDARY OUTCOMES:
Cmax of CJ-16118 (major metabolite of CJ-15314) of single dose of CJ-15314 | Up to 72 hours
Tmax of CJ-16118 (major metabolite of CJ-15314) of single dose of CJ-15314 | Up to 72 hours
AUClast of CJ-16118 (major metabolite of CJ-15314) of single dose of CJ-15314 | Up to 72 hours
AUCinf of CJ-16118 (major metabolite of CJ-15314) of single dose of CJ-15314 | Up to 72 hours
t1/2 of CJ-16118 (major metabolite of CJ-15314) of single dose of CJ-15314 | Up to 72 hours
λz of CJ-16118 (major metabolite of CJ-15314) of single dose of CJ-15314 | Up to 72 hours
Ae of CJ-16118 (major metabolite of CJ-15314) of single dose of CJ-15314 | Up to 72 hours
fe of CJ-16118 (major metabolite of CJ-15314) of single dose of CJ-15314 | Up to 72 hours
Metabolic ratio of CJ-16118 (major metabolite of CJ-15314) of single dose of CJ-15314 | Up to 72 hours
Cmax,ss of CJ-16118 (major metabolite of CJ-15314) of multiple doses of CJ-15314 | Up to 72 hours
Cmin,ss of CJ-16118 (major metabolite of CJ-15314) of multiple doses of CJ-15314 | Up to 72 hours
Cav,ss of CJ-16118 (major metabolite of CJ-15314) of multiple doses of CJ-15314 | Up to 72 hours
Tmax,ss of CJ-16118 (major metabolite of CJ-15314) of multiple doses of CJ-15314 | Up to 72 hours
AUCtau,ss of CJ-16118 (major metabolite of CJ-15314) of multiple doses of CJ-15314 | Up to 72 hours
t1/2 of CJ-16118 (major metabolite of CJ-15314) of multiple doses of CJ-15314 | Up to 72 hours
PTF of CJ-16118 (major metabolite of CJ-15314) of multiple doses of CJ-15314 | Up to 72 hours
Ra of CJ-16118 (major metabolite of CJ-15314) of multiple doses of CJ-15314 | Up to 72 hours
Ae of CJ-16118 (major metabolite of CJ-15314) of multiple doses of CJ-15314 | Up to 72 hours
Metabolic ratio of CJ-16118 (major metabolite of CJ-15314) of multiple doses of CJ-15314 | Up to 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: In-Jin Jang, MD, PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- Seoul National University Hospital, Dept. of Clinical Pharmacology, Seoul, South Korea